CLINICAL TRIAL: NCT04391478
Title: Milrinone Versus Sildenafil in Treatment of PPHN in Neonates
Brief Title: Efficacy and Safety of Milrinone Versus Sildenafil in the Treatment of Neonates With Persistent Pulmonary Hypertension
Acronym: ESMPPHTN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rania Ali El-Farrash (Other)
Responsible Party: Sponsor-Investigator, Rania Ali El-Farrash, assistant professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCT 30
Record Dates: First submitted 2015-10-01; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Persistent Pulmonary Hypertension
MeSH Terms: interventions — Milrinone; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- milrinone (Active Comparator): Milrinone is a phosphodiesterase inhibitor typ3 used in treatment of PPHN. used in dose (0.25 to 0.75 mg/kg/min) intravenous infusion compared with nasogastric sildenafil.
  Interventions: Drug: Milrinone
- sildenafil (Active Comparator): Sildenafil is a phosphodiesterase inhibitor typ 5 used in treatment of PPHN. used in dose (0.2 to 0.5 mg/kg/6h) by nasogastric tube compared with intravenous milrinone infusion.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Milrinone — milrinone lactate, 1mg/ml, for intra venous use only
  Other Names: primacor
  Arms: milrinone
Drug: Sildenafil — 50mg sildenafil citrate/tablet, crushed in water taken by nasogastric tube
  Other Names: Viagra
  Arms: sildenafil

SUMMARY:
Compare the effect of milrinone versus sildenafil in treatment of neonates with persistent pulmonary hypertension.

DETAILED DESCRIPTION:
40 neonates with PPHN, met inclusion criteria, randomly assigned to 2 groups, each includes 20, first group received intravenous milrinone and second group received nasogastric sildenafil. both groups receive other supportive care.

ELIGIBILITY:
Inclusion Criteria:

* gestational age >34 weeks
* postnatal age <10 days

Exclusion Criteria:

* neonates with congenital heart disease
* neonates with congenital diaphragmatic hernia

Ages: 1 Hour to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
efficacy of milrinone versus sildenafil in treatment of PPHN | 6 - 12 months
  effect on oxygenation index

SECONDARY OUTCOMES:
final outcome | 6 - 12 months
  Mortality
Bleeding | 6-12 months
  Bleeding (e.g pulmonary hemorrhage) that is believed to be attributed to medication
Ventilation | 6-12 months
  total duration of mechanical ventilation
Ventilatory settings | 6-12 months
  highest ventilator settings

REFERENCES:
- [Derived] Imam SS, El-Farrash RA, Taha AS, Saleh GA. Milrinone Versus Sildenafil in Treatment of Neonatal Persistent Pulmonary Hypertension: A Randomized Control Trial. J Cardiovasc Pharmacol. 2022 Nov 1;80(5):746-752. doi: 10.1097/FJC.0000000000001332. PMID 35881893